CLINICAL TRIAL: NCT06214559
Title: Prospective Multicentric, Before After Study to Evaluate the Effectiveness and the Safety of a Medical Device in the Treatment of Common Warts and Plantar Warts.
Brief Title: Evaluate the Effectiveness and the Safety of a Medical Device in the Treatment of Common Warts and Plantar Warts.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Footcare Laboratories - Poderm Professional (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23E2007
Record Dates: First submitted 2023-12-28; First posted 2024-01-19 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Warts; Plantar Wart; Common Wart
MeSH Terms: conditions — Warts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serum VERRUPRO (Experimental): To be applied twice a day
  Interventions: Device: Sérum VERRUPRO

INTERVENTIONS:
Device: Sérum VERRUPRO — To be applied twice a day

SUMMARY:
The principal aim of this study is to evaluate the efficacy and the safety of the tested product on common and plantar wart after 35 days of treatment.

For this study, 33 patients presenting at least one common wart on the fingers, back on the hand or a plantar wart of a size between 0.1 and 0.5cm and present since less than 6 months will be included to reach this objective

DETAILED DESCRIPTION:
Warts are the cutaneous manifestations of human papillomavirus (HPV). (1) Cutaneous warts are benign, spontaneously regressing, epithelial tumors differing in clinical morphology depending on the human papilloma virus HPV-types. (2) Warts may exist in different forms given the epithelial surface and HPV type responsible for the infection. Common warts (Verruca vulgaris), plantar warts (Verruca plantaris), flat or planar warts (Verruca plana), and genital warts (Condyloma acuminata) are some of the clinical manifestations of HPV infection. (1) Warts are most common on your hands, feet, and face. (3)

Warts are common worldwide and affect approximately 10% of the population. In school-aged children, the prevalence is as high as 10% to 20% (4). The range of greatest incidence is between 12 and 16 years of age. (1) It is known that nearly two-thirds of warts spontaneously disappear within 24 months. (4)

The majority of warts do not cause symptoms. However, they do cause cosmetic disfigurement and, in a rare patient, may cause localized pain. Plantar warts can be painful because of compression and extensive friction that can lead to bleeding. (4) Once the diagnosis is made, the treatment depends on symptoms, patient preferences, and cost. Even though there are many treatments for warts, none is very effective, and recurrences are common with each of them. (4) This is why, developing a product that is effective against warts seems necessary.

PODERM Professional has developed an innovative wart-treatment formula based on biomimetics. The principal aim of this study is to evaluate the efficacy and the safety of the tested product on common and plantar wart after 35 days of treatment. For this study, 33 patients presenting at least one common wart on the fingers, back on the hand or a plantar wart of a size between 0.1 and 0.5cm and present since less than 6 months will be included to reach this objective.

ELIGIBILITY:
Inclusion Criteria:

Patient having given freely her/his informed, written consent. Patient having a good general health. Age: more than 18 years. Patient cooperative and aware of the device's modalities of use and the necessity and duration of the controls so that perfect adhesion to the protocol can be expected.

Patient being psychologically able to understand information and to give his/her consent.

Patient presenting at least 1 common wart, present since less than 6 months, on the fingers, back of the hands (60% of patients) and/or at least 1 plantar wart (40% of patients).

Patient presenting wart of a size between 0,1 and 0,5 cm. Women of childbearing potential should use an accepted contraceptive regimen (at the Investigator's discretion) since at least 12 weeks before the beginning of the study and during all the study.

Exclusion Criteria:

For plantar wart: wart on the point of support. Wart with keratosis. Wart in mosaic. Pregnant or nursing woman or planning a pregnancy during the investigation. Patient considered by the investigator likely to be non-compliant with the protocol.

Patient enrolled in another clinical trial during the test period. Patient having a known allergy or hypersensitivity to one of the constituents of the tested products.

Patient with a condition or receiving a medication which, in the investigator's judgment, put the patient at undue risk.

Patient suffering from serious or progressive diseases (to investigator's discretion) such as uncontrolled diabetes, peripheral circulatory disease, immunocompromised patient HIV, psoriasis, lichen planus, immunosuppressive pathology, chronic venous insufficiency, Peripheral Arterial Obstructive Disease, delay or lack of ungual growth … Patient with cutaneous pathology on studied zone other than warts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Tunisia (2):
  - L'Activité Privée Complémentaire (APC) Habib Thameur hospital, Tunis
  - Private practice, Tunis

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in two private prictise in Tunisia from 19.02.2024 to 16.07.2024
Pre-assignment Details: Not applicable. No enrolled patient were excluded from the study before groups assignments
Period: Overall Study
Arm/Group | Serum VERRUPRO
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Serum VERRUPRO
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.15 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Tunisia | 33

OUTCOME MEASURES:

1. Primary Outcome: Diameter of the Wart
Description: Clinical examination performed by the investigator to evaluate the diameter of the wart at D0 and 35 days after treatment.
  The effect of the product on clinical parameters will be evaluated by comparing the mean diameter before and after treatment.
Time Frame: Day 0, Day 35
Population: On ITT population
Measure: Mean (Standard Error); unit: cm
Arm/Group | Serum VERRUPRO
Number analyzed (Participants) | 33
cm | -0.12 (0.14)

2. Secondary Outcome: Global Improvement of the Wart
Description: The global improvement of the wart will be assessed by the investigator after 35 days of treatment.
Time Frame: Day 35
Population: On per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Serum VERRUPRO
Number analyzed (Participants) | 32
Participants
  Beginning of improvement | 15
  Significant improvement | 12
  Total recovery | 4
  No change | 1

3. Secondary Outcome: Roughness of the Wart
Description: The effect of the product on these clinical parameters will be evaluated by a comparison before and after treatment. This outcome was measured using a scale from 0 (No roughness) to 5 (very severe roughness).
Time Frame: Day 0, Day 35
Population: On per protocol population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Serum VERRUPRO
Number analyzed (Participants) | 32
score on a scale | -1.4 (1.0)

4. Secondary Outcome: Thickness of the Wart
Description: The effect of the product on these clinical parameters will be evaluated by a comparison before and after treatment. This outcome was measured using a scale form 0 (no tickness) to 4(Very severe)
Time Frame: Day 0, Day 35
Population: On per protocol population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Serum VERRUPRO
Number analyzed (Participants) | 32
score on a scale | -1.5 (0.8)

5. Secondary Outcome: Number of Dermal Papillae
Description: The effect of the product on these clinical parameters will be evaluated by a comparison before and after treatment.
Time Frame: Day 0, Day 35
Population: On per protocol population
Measure: Mean (Standard Deviation); unit: number of dermal papillae
Arm/Group | Serum VERRUPRO
Number analyzed (Participants) | 32
number of dermal papillae | -4.1 (3.8)

6. Secondary Outcome: Number of Participants Who Participated in Photography Session
Description: Illustration of the effectiveness of Sérum VERRUPRO® on the skin aspect before and after the treatment with photographs. A standardized photographs was taken at D0 an D35 in order to illustrate the effect of the product. No data were measured on these pictures.
  Number of Participants Who Participated in Photography Session
Time Frame: Day 0, Day 35
Population: Only photographs for illustration, no data analysed. Number of Participants Who Participated in Photography Session
Measure: Count of Participants; unit: Participants
Arm/Group | Serum VERRUPRO
Number analyzed (Participants) | 32
Participants | 32

7. Secondary Outcome: Patient Evaluation
Description: Analysis of the answers to the patient questionnaire regarding effectiveness, tolerance, and acceptability of the investigational device 35 days after treatment.
Time Frame: Day 35
Population: On per protocol population, are you globally statisfied with the product
Measure: Count of Participants; unit: Participants
Arm/Group | Serum VERRUPRO
Number analyzed (Participants) | 32
Participants
  totally agree | 8
  agree | 9
  neutral | 11
  disagree | 4
  totally disagree | 0

8. Secondary Outcome: Adverse Event
Description: Products safety will be assessed by collection of Adverse Events (AEs) throughout the study. AEs will be summarized and tabulated by severity, causality, action taken and outcome, using descriptive statistics.
Time Frame: Day 0, Day 35
Population: No adverse event during the study
Measure: Count of Participants; unit: Participants
Arm/Group | Serum VERRUPRO
Number analyzed (Participants) | 33
Participants | 0

9. Secondary Outcome: Product Tolerance
Description: Product tolerance will be assessed by the investigator at D0 (before the product use) and D35 by a clinical examination.
Time Frame: Day 0, Day 35
Population: on per protocol population, evaluation of local tolerance on redness / edema / Desquamation and dryness. here is presented redness at D35
Measure: Count of Participants; unit: Participants
Arm/Group | Serum VERRUPRO
Number analyzed (Participants) | 32
Participants
  None | 18
  Very mild | 9
  Mild | 3
  Moderate | 1
  Severe | 1

ADVERSE EVENTS:
Time Frame: 35 days
Description: No adverse event occured during the study. All adverse evnet were monitored during the study
Arm/Group | Serum VERRUPRO
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT06214559/Prot_SAP_000.pdf